CLINICAL TRIAL: NCT01451294
Title: The Effect of Phenylephrine Versus Ephedrine on Cerebral Perfusion During Carotid Endarterectomy
Brief Title: Effect of Blood Pressure on rSO2 in Carotid Endarterectomy (CEA)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: G.J. de Borst (Other)
Responsible Party: Sponsor-Investigator, G.J. de Borst, Vascular surgeon; Head of cerebrovascular surgical programme., UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11-195
Record Dates: First submitted 2011-09-22; First posted 2011-10-13 (Estimated); Last update posted 2011-10-13 (Estimated); Status verified 2011-10

CONDITIONS: Intra-operative Hypotension; Carotid Stenosis
Keywords: Cerebral autoregulation
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Ephedrine (Active Comparator)
  Interventions: Drug: Administration of ephedrine
- Phenylephrine (Active Comparator)
  Interventions: Drug: Administration of phenylephrine

INTERVENTIONS:
Drug: Administration of phenylephrine — Phenylephrine: 50-100µg
  Arms: Phenylephrine
Drug: Administration of ephedrine — Ephedrine: 5- 10 mg
  Arms: Ephedrine

SUMMARY:
Carotid endarterectomy (CEA) is the recommended treatment for symptomatic high degree stenosis of the internal carotid artery (ICA). ICA obstruction is often associated with an impaired cerebral autoregulation, implicating that cerebral perfusion pressure becomes dependent on systemic blood pressure. Therefore, to maintain cerebral perfusion pressure in this type of patients intraoperative hypotension needs to be avoided. Different short-acting agents such as phenylephrine, (a drug with vasoconstrictive properties), or ephedrine (a drug with vasoconstrictive properties combined with an increase in heart rate) can be used to correct intra-operative hypotension. In healthy subjects these agents affect the cerebral perfusion differently despite an identical effect on the systemic blood pressure. Cerebral perfusion decreases after phenylephrine administration while it is preserved after the use of ephedrine. The optimal agent for correcting hypotension in CEA patients, and thus in a situation of an impaired cerebral autoregulation, is unknown.

Therefore, the investigators propose to perform a prospective study observing the effect of phenylephrine and ephedrine on cerebral perfusion to make a recommendation regarding the use of either phenylephrine or ephedrine during CEA.

ELIGIBILITY:
Inclusion criteria:

1. All patients undergoing CEA in the University Medical Centre Utrecht and having an appropriate temporal bone window for reliable perioperative TCD monitoring could be included.
2. All patients must have given written informed consent.

Exclusion criteria:

1. Not having a temporal bone window appropriate for TCD measurement
2. Not willing to give informed consent.
3. If the effect on BP of the given agents is insufficient (if relative hypotension persists five minutes after administration).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
cerebral perfusion (rSO2) measured using Near Infrared Spectroscopy | (day 1) Monitoring will take place only on the day of operation. No further follow-up. Timeframe is 1 day.
  A continuous measurement during surgery will be performed. However for further analysis only a short time frame will be used.

SECONDARY OUTCOMES:
Blood velocity (Vmca) measured using transcranial Doppler | Within 18 months in consecutive patients undergoing carotid endarterectomy. Endpoints will only be assessed during actual surgery (approximately 90 minutes in total) no data will be assessed during follow-up.
  A continuous measurement during surgery will be performed. However for further analysis only a short time frame will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Gert Jan de Borst, MD, PhD, Study Director — UMC Utrecht, The Netherlands; Claire Pennekamp, MD, Principal Investigator — UMC Utrecht, The Netherlands
Locations (1):
- University Medical Center Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Background] Nissen P, Brassard P, Jorgensen TB, Secher NH. Phenylephrine but not ephedrine reduces frontal lobe oxygenation following anesthesia-induced hypotension. Neurocrit Care. 2010 Feb;12(1):17-23. doi: 10.1007/s12028-009-9313-x. PMID 19957053
- [Derived] Fassaert LMM, de Borst GJ, Pennekamp CWA, Specken-Welleweerd JC, Moll FL, van Klei WA, Immink RV. Effect of Phenylephrine and Ephedrine on Cerebral (Tissue) Oxygen Saturation During Carotid Endarterectomy (PEPPER): A Randomized Controlled Trial. Neurocrit Care. 2019 Dec;31(3):514-525. doi: 10.1007/s12028-019-00749-w. PMID 31190322
- [Derived] Heusdens JF, Lof S, Pennekamp CW, Specken-Welleweerd JC, de Borst GJ, van Klei WA, van Wolfswinkel L, Immink RV. Validation of non-invasive arterial pressure monitoring during carotid endarterectomy. Br J Anaesth. 2016 Sep;117(3):316-23. doi: 10.1093/bja/aew268. PMID 27543526
- [Derived] Pennekamp CW, Immink RV, Buhre WF, Moll FL, de Borst GJ. Phenylephrine versus ephedrine on cerebral perfusion during carotid endarterectomy (PEPPER): study protocol for a randomized controlled trial. Trials. 2013 Feb 14;14:43. doi: 10.1186/1745-6215-14-43. PMID 23410186